CLINICAL TRIAL: NCT01153321
Title: A Single-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Phase IIa Study to Investigate the Effects of 100mg AZD2423 as an Oral Tablet in Subjects With Mild COPD Following Segmental Endobronchial LPS Instillation
Brief Title: Investigation of the Effect of Oral Treatment With 100 mg AZD2423 in Subjects With Mild Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3320C00001; 2010-020141-26 (EudraCT Number)
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Disease
Keywords: Respiratory disease; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral treatment
  Interventions: Drug: AZD2423
- 2 (Placebo Comparator): Oral treatment
  Interventions: Drug: AZD2423 Placebo

INTERVENTIONS:
Drug: AZD2423 — 100mg Oral dose od
  Arms: 1
Drug: AZD2423 Placebo — Oral dose od
  Arms: 2

SUMMARY:
The purpose of the study is to find out if AZD2423 can reduce inflammation in the lungs of patients with mild COPD.

ELIGIBILITY:
Inclusion Criteria:

* Only women of non-child bearing potential are included in the study i.e. women who are permanently or surgically sterilised or post menopausal.
* ≥ 40 years of age at Visit 1
* Clinical diagnosis of COPD (GOLD stage 1)
* FEV1 ≥ 80% of the predicted normal post-bronchodilator at Visit 1 (GOLD stage 1)
* FEV1/FVC <70% post-bronchodilator at Visit 1 (GOLD stage 1)

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk or influence the way the drug works
* Any clinically relevant abnormal findings in physical examination, blood or urine test results, vital signs or ECG at Visit 1 that may put the subject at risk during the study, affect their ability or take part or influence the results of the study
* A past history or current indication of renal (kidney) failure
* Subjects at risk of active tuberculosis or of disease reactivation
* Subjects who have had any clinically significant illness within 4 weeks before Visit 2 (start of treatment)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Larsson, Study Director — AstraZeneca R&D
Locations (1):
- Research Site, Hanover, Hannover, Germany

REFERENCES:
- See also: D3320C00001 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=206&filename=CSR-D3320C00001.pdf
- See also: D3320C00001 CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=206&filename=D3320C00001.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single centre study conducted at a medical research centre in Germany. The first patient was enrolled on 01 October 2010 and the last patient last visit was on 28 July 2011.
  A total of 71 subjects were enrolled to get 44 subjects that fulfilled the inclusion criterions.
Groups:
- AZD2423: Two 50 mg AZD2423 tablets, once daily
- Placebo: Placebo to match AZD2423 tablets, once daily
Period: Overall Study
Arm/Group | AZD2423 | Placebo
Started | 22 | 22
Completed | 21 | 19
Not Completed | 1 | 3
Not completed — Development of study withdrawal criteria | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2423 | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (7.6) | 54.1 (8.1) | 53 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 20 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Absolute Monocyte Count in BAL Post-LPS Challenge
Description: Monocyte count in BAL post-LPS challenge (Day 11)
Time Frame: Day 11
Population: Thirty-nine patients were included in the efficacy analysis set. Five patients were excluded because they did not have sufficient data to be included in the primary outcome analysis. Four discontinued and one did not complete LPS challenge
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 398 (1.276) | 514.4 (1.284)

2. Secondary Outcome: Total Neutrophils in Biopsy Sample (Post-LPS Challenge)
Description: Pre-challenge = Day 11. Biopsies taken from left lingula. Cells counted in subepithelium.
Time Frame: Day 11
Population: Thirty-nine patients were included in the efficacy analysis set. Five patients were excluded because they did not have sufficient data to be included in the primary outcome analysis. Four discontinued and one did not complete LPS challenge. Six patients had missing observations.
Measure: Least Squares Mean (Standard Error); unit: cells/mm^2
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 18 | 15
cells/mm^2 | 20.7 (1.218) | 34.04 (1.258)

3. Secondary Outcome: Total Macrophages in Biopsy Sample (Post-LPS Challenge)
Description: Post-LPS challenge data (Day 11). Post-LPS challenge biopsies taken from right middle lobe. Cells counted in subepithelium.
Time Frame: Day 11
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cells/mm^2
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 18 | 15
cells/mm^2 | 28.44 (1.233) | 41.17 (1.274)

4. Secondary Outcome: CD45+ in Biopsy Sample (Post-LPS Challenge)
Description: as for outcome 3
Time Frame: Day 11
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cells/mm^2
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 18 | 15
cells/mm^2 | 200.7 (1.133) | 203.2 (1.156)

5. Secondary Outcome: CD3+ in Biopsy Sample (Post-LPS Challenge)
Description: as for outcome 3
Time Frame: Day 11
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cells/mm^2
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 18 | 15
cells/mm^2 | 71.84 (1.212) | 81.1 (1.249)

6. Secondary Outcome: Biopsy PAS Reaction Grade (Post-LPS Challenge)
Description: Biopsies stained using PAS method. Graded on subjective scale (1=normal; 2=PAS positive cell hypertrophy; 3=PAS positive cell hyperplasia; 4=Metaplasia with PAS positive cells throughout mucosa; 5=Metaplasia and/or squamous plates with loss of PAS positive cells).
Time Frame: Day 11
Population: Thirty-nine patients were included in the efficacy analysis set. Five patients were excluded because they did not have sufficient data to be included in the primary outcome analysis. Four discontinued and one did not complete LPS challenge. Thirteen patients had missing observations.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 14 | 12
Units on a scale | 2.55 (0.415) | 2.5 (0.615)

7. Secondary Outcome: Biopsy Epithelium Grade (Post-LPS Challenge)
Description: Biopsies (from right middle lobe) were assessed for routine histopathology. Epithelial morphology was graded on subjective scale from 1 to 5. 1=normal; 2=PAS positive cell hypertrophy; 3=PAS positive cell hyperplasia; 4=Metaplasia with PAS positive cells throughout mucosa; 5=Metaplasia and/or squamous plates with loss of PAS positive cells
Time Frame: Day 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 14 | 12
Units on a scale | 2.32 (0.32) | 2.29 (0.475)

8. Secondary Outcome: Eosinophils in BAL (Post-LPS Challenge)
Description: Post-LPS challenge eosinophil differential in BAL. LPS challenge and post-challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: Thirty-nine patients were included in the efficacy analysis set. Five patients were excluded because they did not have sufficient data to be included in the primary outcome analysis. Four discontinued and one did not complete LPS challenge. Five patients had missing observations.
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 18 | 16
x10^4 cells/mL | 28.15 (1.264) | 61.35 (1.338)

9. Secondary Outcome: Lymphocytes in BAL (Post-LPS Challenge)
Description: Post-LPS challenge lymphocyte differential in BAL. LPS challenge and post-challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 129.7 (1.242) | 161.7 (1.257)

10. Secondary Outcome: Neutrophils in BAL (Post-LPS Challenge)
Description: Post-LPS challenge neutrophil differential in BAL. LPS challenge and post-challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 2063 (1.3) | 1890 (1.319)

11. Secondary Outcome: Macrophages in BAL (Post-LPS Challenge)
Description: Post-LPS challenge macrophage differential in BAL. LPS challenge and post-challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 771.1 (1.181) | 917.7 (1.186)

12. Secondary Outcome: TNF α Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge TNF α concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: Thirty-nine patients were included in the efficacy analysis set. Five patients were excluded because they did not have sufficient data to be included in the primary outcome analysis. Four discontinued and one did not complete LPS challenge. One patient had missing observations.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 18
pg/mL | 2.16 (1.134) | 3.11 (1.142)

13. Secondary Outcome: CCL2 Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge CCL2 concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 18
pg/mL | 82.47 (1.128) | 46.25 (1.136)

14. Secondary Outcome: IL-1β Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge IL-1β concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 18
pg/mL | 0.91 (1.15) | 1.05 (1.159)

15. Secondary Outcome: IL-6 Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge IL-6 concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 18
pg/mL | 13.97 (1.213) | 19.76 (1.226)

16. Secondary Outcome: IL-8 Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge IL 8 concentration in BAL. LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 18
pg/mL | 182.5 (1.114) | 207.8 (1.121)

17. Secondary Outcome: RANTES Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge RANTES concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 18
pg/mL | 3.89 (1.16) | 4.82 (1.169)

18. Secondary Outcome: SP-D Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge SP-D concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 19 | 19
ng/mL | 637.3 (1.081) | 799.1 (1.079)

19. Secondary Outcome: SAA Concentration in Blood (Pre-LPS Challenge)
Description: SAA concentration in blood pre-LPS challenge (Day 10).
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
ng/mL | 2312 (1.168) | 2510 (1.173)

20. Secondary Outcome: SAA Concentration in Blood (Post-LPS Challenge)
Description: SAA concentration in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
ng/mL | 18615 (1.201) | 16312 (1.207)

21. Secondary Outcome: CCL2 Concentration in Blood (Pre-LPS Challenge)
Description: CCL2 concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 1212 (1.041) | 323.4 (1.042)

22. Secondary Outcome: CCL2 Concentration in Blood (Post-LPS Challenge)
Description: CCL2 concentration in blood post-LPS challenge (Day 11).
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 1182 (1.061) | 292.9 (1.063)

23. Secondary Outcome: IL-1β Concentration in Blood (Pre-LPS Challenge)
Description: IL-1β concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 1.26 (1.055) | 1.14 (1.056)

24. Secondary Outcome: IL-1β Concentration in Blood (Post-LPS Challenge)
Description: IL-1β concentration in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 1.12 (1.017) | 1.12 (1.017)

25. Secondary Outcome: IL-6 Concentration in Blood (Pre-LPS Challenge)
Description: IL-6 concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 2.61 (1.087) | 2.55 (1.09)

26. Secondary Outcome: IL-6 Concentration in Blood (Post-LPS Challenge)
Description: IL-6 concentration in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 4.41 (1.215) | 2.87 (1.221)

27. Secondary Outcome: IL-8 Concentration in Blood (Pre-LPS Challenge)
Description: IL-8 concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 8.37 (1.059) | 9.47 (1.061)

28. Secondary Outcome: IL-8 Concentration in Blood (Post-LPS Challenge)
Description: IL-8 concentration in blood post-LPS challenge (Day 11)
Time Frame: day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 12.14 (1.193) | 8.85 (1.199)

29. Secondary Outcome: TNF-α Concentration in Blood (Pre-LPS Challenge)
Description: TNF-α concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 13.07 (1.095) | 12.55 (1.097)

30. Secondary Outcome: TNF-α Concentration in Blood (Post-LPS Challenge)
Description: TNF-α concentration in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 12.11 (1.09) | 11.19 (1.092)

31. Secondary Outcome: SP-D Concentration in Blood (Pre-LPS Challenge)
Description: SP-D concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
ng/mL | 201.8 (1.043) | 181.6 (1.044)

32. Secondary Outcome: SP-D Concentration in Blood (Post-LPS Challenge)
Description: SP-D concentration in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
ng/mL | 198.8 (1.041) | 185.6 (1.042)

33. Secondary Outcome: CC16 Concentration in Blood (Pre-LPS Challenge)
Description: CC16 concentration in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: Thirty-nine patients were included in the efficacy analysis set. Five patients were excluded because they did not have sufficient data to be included in the primary outcome analysis. Four discontinued and one did not complete LPS challenge. Three patients had missing observations.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 19 | 17
ng/mL | 123.2 (1.034) | 125.4 (1.037)

34. Secondary Outcome: CC16 Concentration in Blood (Post-LPS Challenge)
Description: CC16 concentration in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 19 | 15
ng/mL | 113.7 (1.039) | 121.6 (1.044)

35. Secondary Outcome: Basophils in Blood (Pre-LPS Challenge)
Description: Basophils in blood pre-LPS challenge (Day 10)
Time Frame: day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 2.87 (1.106) | 3.06 (1.106)

36. Secondary Outcome: Basophils in Blood (Post-LPS Challenge)
Description: Basophils in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 2.68 (1.145) | 3.02 (1.15)

37. Secondary Outcome: Eosinophils in Blood (Pre-LPS Challenge)
Description: Eosinophils in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 17.19 (1.161) | 17.32 (1.161)

38. Secondary Outcome: Eosinophils in Blood (Post-LPS Challenge)
Description: Eosinophils in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 15.7 (1.092) | 19.8 (1.092)

39. Secondary Outcome: Lymphocytes in Blood (Pre-LPS Challenge)
Description: Lymphocytes in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 226.6 (1.035) | 215.2 (1.035)

40. Secondary Outcome: Lymphocytes in Blood (Post-LPS Challenge)
Description: Lymphocytes in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 215.7 (1.043) | 198.8 (1.043)

41. Secondary Outcome: Monocytes in Blood (Pre-LPS Challenge)
Description: Monocytes in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 45.17 (1.13) | 51.11 (1.13)

42. Secondary Outcome: Monocytes in Blood (Post-LPS Challenge)
Description: Monocytes in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 51.99 (1.053) | 63.33 (1.053)

43. Secondary Outcome: Neutrophils in Blood (Pre-LPS Challenge)
Description: Neutrophils in blood pre-LPS challenge (Day 10)
Time Frame: Day 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 461.6 (1.055) | 464.4 (1.055)

44. Secondary Outcome: Neutrophils in Blood (Post-LPS Challenge)
Description: Neutrophils in blood post-LPS challenge (Day 11)
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: x10^4 cells/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
x10^4 cells/mL | 552.4 (1.083) | 514.7 (1.083)

45. Secondary Outcome: Maximum Plasma Concentration (Cmax) of AZD2423 at Steady State
Description: Steady state pharmacokinetic (PK) profile measured on Day 10
Time Frame: Day 10 pre-dose, 20 and 40 minutes post-dose, 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: All 22 patients who received AZD2423 provided at least one plasma sample and were included in the PK analysis although only 21 patients were included in the evaluation of PK at day 10, one patient had been discontinued due to an AE.
Measure: Geometric Mean (Full Range); unit: nmol/L
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 21 | 0
nmol/L | 228.77 [94.3 to 655.0] |

46. Secondary Outcome: Time to Cmax (Tmax) of AZD2423 at Steady State
Description: Steady state PK profile measured on Day 10
Time Frame: Day 10 pre-dose, 20 and 40 minutes post-dose, 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 45
Measure: Median (Full Range); unit: hours
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 21 | 0
hours | 0.3 [0.3 to 4.0] |

47. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 24 Hours (AUC(0-24)) of AZD2423 at Steady State
Description: Steady state PK profile measured on Day 10
Time Frame: Day 10 pre-dose, 20 and 40 minutes post-dose, 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 45
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 21 | 0
nmol*h/L | 1454.14 [872.7 to 2259.0] |

48. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 8 Hours (AUC(0-8)) of AZD2423 at Steady State
Description: Steady state PK profile measured on Day 10
Time Frame: Day 10 pre-dose, 20 and 40 minutes post-dose, 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 45
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 21 | 0
nmol*h/L | 801.25 [488.5 to 1182.9] |

49. Secondary Outcome: Number of Participants With Clinically Relevant Treatment-related Changes in Laboratory Variables Other Than Monocytes
Time Frame: up to 47 days (visit 1 to visit 6)
Measure: Number; unit: Participants
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

50. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Vital Signs
Time Frame: up to 47 days (visit 1 to visit 6)
Measure: Number; unit: Participants
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

51. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Electrocardiogram (ECG) Variables
Time Frame: up to 47 days (visit 1 to visit 6)
Measure: Number; unit: Participants
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

52. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Physical Examination
Time Frame: up to 47 days (visit 1 to visit 6)
Measure: Number; unit: Participants
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

53. Secondary Outcome: Number of Participants With Treatment-related or Clinically Relevant Changes in Spirometry (Forced Expiratory Volume in 1 Second [FEV1], Forced Vital Capacity [FVC] Pre-bronchodilator)
Time Frame: up to 47 days (visit 1 to visit 6)
Measure: Number; unit: Participants
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

54. Secondary Outcome: CC16 Concentration in BAL (Post-LPS Challenge)
Description: Post-LPS challenge CC16 concentration in BAL (Day 11). LPS challenge and post-LPS challenge BAL conducted at right middle lobe.
Time Frame: Day 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | AZD2423 | Placebo
Number analyzed (Participants) | 20 | 19
ng/mL | 2256 (1.132) | 2589 (1.136)

ADVERSE EVENTS:
Arm/Group | AZD2423 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 3/22
Other Adverse Events (participants affected / at risk) | 10/22 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD2423 100 mg (N=22) | Placebo (N=22)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD2423 100 mg (N=22) | Placebo (N=22)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 2 (3)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
FATIGUE (General disorders) | 0 (0) | 2 (2)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2) | 5 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
VASOMOTOR RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institutions or Investigators were permitted to publish or present the study results from their site (or the overall results), providing the article or presentation was submitted to and approved by AstraZeneca beforehand.